CLINICAL TRIAL: NCT06276829
Title: A Convenient Parameter for Predicting Behçet's Disease Severity: Lactate Dehydrogenase/Albumin Ratio
Brief Title: Behçet and LDH/Albumin
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erdal Pala, Department of Skin and Venereal Diseases, Ataturk University
Other Study IDs: 02.05.2023/291
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Behcet's Disease; Albumin; Lactate Dehydrogenase; Disease Severity
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behçet's Disease
  Interventions: Diagnostic Test: LDH/albumin ratio
- healthy individuals
  Interventions: Diagnostic Test: LDH/albumin ratio

INTERVENTIONS:
Diagnostic Test: LDH/albumin ratio — LDH/Albumin ratios of patient and control groups were recorded.

SUMMARY:
ABSTRACT Objective: To investigate whether the lactate dehydrogenase to albumin ratio can be used as a parameter to determine disease severity in Behçet's disease, an inflammatory disease, by comparing it to healthy controls.

Patients and Methods: In this retrospective cohort study, patients with Behçet's disease aged 18-69 years who presented to the outpatient clinic between February 2020 and April 2023 and healthy individuals of similar age and gender were enrolled. LDH, albumin levels, and LDH/albumin ratio of both groups were compared. Clinical findings and characteristics of Behçet's patients and disease severity were recorded and analyzed in relation to LDH/albumin ratio.

ELIGIBILITY:
Inclusion Criteria:

Patients with Behçet's disease aged 18-69

Exclusion Criteria:

* younger than 18 years or older than 69 years, pregnant and lactating patients, patients with acute infection on admission or nutritional problems, symptomatic gastrointestinal symptoms, malignancy, hepatitis or liver disease were excluded.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 349 subjects, including 160 patients with Behçet's disease and 189 healthy controls
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
LDH/albumin ratio | February 2020 and April 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Erdal Pala, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pala E, Bayraktar M. Lactate dehydrogenase to albumin ratio as a convenient parameter for predicting the severity of Behcet disease: a cross-sectional study. BMC Immunol. 2026 Jan 7;27(1):1. doi: 10.1186/s12865-025-00706-7. PMID 41501648